CLINICAL TRIAL: NCT02136420
Title: Countermeasures to Reduce Sensorimotor Impairment and Space Motion Sickness Resulting From Altered Gravity Levels
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Faisal_Karmali@MEEI.HARVARD.EDU (Other)
Collaborators: National Space Biomedical Research Institute (Other); Massachusetts Institute of Technology (Other)
Responsible Party: Sponsor-Investigator, Faisal_Karmali@MEEI.HARVARD.EDU, Primary Investigator, Massachusetts Eye and Ear Infirmary
Organization: Massachusetts Eye and Ear Infirmary (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 497997
Record Dates: First submitted 2014-04-30; First posted 2014-05-13 (Estimated); Results first posted 2018-01-08 (Actual); Last update posted 2018-01-08 (Actual); Status verified 2017-12

CONDITIONS: Vestibular
MeSH Terms: interventions — Promethazine; Starch

STUDY DESIGN:
Intervention Model Description: The design includes three separate studies:
  1. Arm 9&10 follows a crossover design. These results were reported in Diaz-Artiles et al 2017.
  2. Arms 1-4 are a separate study which follow a factorial design, with arm 2 serving as the placebo, arms 1 and 3 assessing the effects of two separate interventions and arm 4 assessing the effect of two combined interventions.
  3. Arms 5-8 are a separate study which follow a factorial design, with arm 6 serving as the placebo, arms 5 and 7 assessing the effects of two separate interventions and arm 8 assessing the effect of two combined interventions.
Who Masked: Participant, Investigator
Masking Description: Double masking applies to arms 9&10. Other arms use participant masking only.
Oversight: Data Monitoring Committee: No

ARMS (10):
- Tilt perception, Training, placebo (Experimental): placebo
  Interventions: Behavioral: Hyper gravity training; Drug: Placebo
- Tilt perception, No training, placebo (Placebo Comparator): subject does test with no hypergravity training and placebo drug only
  Interventions: Drug: Placebo; Behavioral: No hypergravity training
- Tilt perception, Training, promethazine (Experimental): promethazine 25 mg, one time 120 minutes prior to experiment
  Interventions: Drug: Promethazine; Behavioral: Hyper gravity training
- Tilt perception,No training,promethazine (Experimental): promethazine 25 mg, one time 120 minutes prior to experiment. No hypergravity training
  Interventions: Drug: Promethazine; Behavioral: No hypergravity training
- Manual Control, Training, placebo (Experimental): placebo
  Interventions: Behavioral: Hyper gravity training; Drug: Placebo
- Manual Control, No training, placebo (Placebo Comparator): subject does test with no hyper gravity training and placebo drug only
  Interventions: Drug: Placebo; Behavioral: No hypergravity training
- Manual Control, Training, promethazine (Experimental): promethazine 25 mg, one time 120 minutes prior to experiment
  Interventions: Drug: Promethazine; Behavioral: Hyper gravity training
- Manual Control,No training,promethazine (Experimental): promethazine 25 mg, one time 120 minutes prior to experiment
  Interventions: Drug: Promethazine; Behavioral: No hypergravity training
- Perceptual thresholds,drug then placebo (Experimental): Subjects undergo perceptual motion threshold tests to determine the smallest motion they can reliably sense for yaw rotation, interaural translation and roll tilt. Each subject is tested twice, once with promethazine then once with placebo, separated by >4 days.
  This arm corresponds to results published in Diaz-Artiles et al 2017.
  Interventions: Drug: Promethazine; Drug: Placebo
- Perceptual thresholds,placebo then drug (Experimental): Subjects undergo perceptual motion threshold tests to determine the smallest motion they can reliably sense for yaw rotation, interaural translation and roll tilt. Each subject is tested twice, once with placebo then once with promethazine, separated by >4 days.
  This arm corresponds to results published in Diaz-Artiles et al 2017.
  Interventions: Drug: Promethazine; Drug: Placebo

INTERVENTIONS:
Drug: Promethazine — Subject receives promethazine
  Other Names: Phenergan
  Arms: Manual Control, Training, promethazine; Manual Control,No training,promethazine; Perceptual thresholds,drug then placebo; Perceptual thresholds,placebo then drug; Tilt perception, Training, promethazine; Tilt perception,No training,promethazine
Behavioral: Hyper gravity training — Subject receives hypergravity training before testing
  Arms: Manual Control, Training, placebo; Manual Control, Training, promethazine; Tilt perception, Training, placebo; Tilt perception, Training, promethazine
Drug: Placebo — Placebo
  Other Names: corn starch
  Arms: Manual Control, No training, placebo; Manual Control, Training, placebo; Perceptual thresholds,drug then placebo; Perceptual thresholds,placebo then drug; Tilt perception, No training, placebo; Tilt perception, Training, placebo
Behavioral: No hypergravity training — Subjects do not receive normal Earth gravity
  Arms: Manual Control, No training, placebo; Manual Control,No training,promethazine; Tilt perception, No training, placebo; Tilt perception,No training,promethazine

SUMMARY:
The investigators will study adaptation of motion perception and manual control in altered gravity, including the effects of a drug (promethazine). The investigators will also study whether promethazine affects motion perceptual thresholds.

DETAILED DESCRIPTION:
Adaptation to altered gravity has been of concern from the earliest reports of space motion sickness, through the Apollo exploration era, and into current planning of exploration missions. The proposed research program takes a new approach which could lead to an effective, practical and acceptable protocol for preadapting astronauts to space flight. By using the gravito-inertial alterations possible with centrifugation in different body orientations the investigators will quantify an individual's sensory adaptation capability and use it to predict and to minimize the consequences of movement in any other gravity environment - eventually including weightlessness. The investigators will also study whether a drug (promethazine) affects motion perception and motion sickness.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be in general good health

Exclusion Criteria:

* Anyone who is not generally in good general health does not qualify
* Cardiovascular disease
* Severe diabetes
* Respiratory condition (e.g. asthma or emphysema)
* Narrow angle glaucoma
* Prostatic hypertrophy
* Gastrointestinal disorders

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2014-06; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Faisal Karmali, Ph.D., Principal Investigator — Massachusetts Eye and Ear Infirmary
Locations (1):
- Massachusetts Eye and Ear Infirmary, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Diaz-Artiles A, Priesol AJ, Clark TK, Sherwood DP, Oman CM, Young LR, Karmali F. The Impact of Oral Promethazine on Human Whole-Body Motion Perceptual Thresholds. J Assoc Res Otolaryngol. 2017 Aug;18(4):581-590. doi: 10.1007/s10162-017-0622-z. Epub 2017 Apr 24. PMID 28439720

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Tilt Perception, Training, Placebo | Tilt Perception, No Training, Placebo | Tilt Perception, Training, Promethazine | Tilt Perception,No Training,Promethazine | Manual Control, Training, Placebo | Manual Control, No Training, Placebo | Manual Control, Training, Promethazine | Manual Control,No Training,Promethazine | Perceptual Thresholds,Drug Then Placebo | Perceptual Thresholds,Placebo Then Drug
Started | 10 | 0 | 0 | 0 | 10 | 0 | 0 | 0 | 5 | 5
Completed | 9 | 0 | 0 | 0 | 10 | 0 | 0 | 0 | 5 | 5
Not Completed | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Perceptual Thresholds,Drug Then Placebo: Subjects undergo perceptual motion threshold tests to determine the smallest motion they can reliably sense for yaw rotation, interaural translation and roll tilt. Each subject is tested twice, once with promethazine then once with placebo, separated by >4 days.
  Promethazine: Subject receives promethazine
  Placebo: Placebo
- Perceptual Thresholds,Placebo Then Drug: Subjects undergo perceptual motion threshold tests to determine the smallest motion they can reliably sense for yaw rotation, interaural translation and roll tilt. Each subject is tested twice, once with placebo then once with promethazine, separated by >4 days.
  Promethazine: Subject receives promethazine
  Placebo: Placebo
- Total: Total of all reporting groups
Arm/Group | Tilt Perception, Training, Placebo | Manual Control, Training, Placebo | Perceptual Thresholds,Drug Then Placebo | Perceptual Thresholds,Placebo Then Drug | Total
Number analyzed (Participants) | 10 | 10 | 5 | 5 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.3 (6.4) | 28.0 (6.3) | 27.4 (4.2) | 24.8 (2.9) | 27.6 (4.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 6 | 1 | 2 | 13
  Male | 6 | 4 | 4 | 3 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 1 | 1 | 4
  Not Hispanic or Latino | 9 | 9 | 4 | 4 | 26
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 3 | 3 | 0 | 0 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 1 | 0 | 2
  White | 6 | 7 | 4 | 3 | 20
  More than one race | 0 | 0 | 0 | 2 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Roll Tilt Perception After Exposure to Hypogravity
Description: Note that this applies to arms 1-4 only.
  Subjects sat on a chair on a moving platform on top of a centrifuge that created an artificial gravity environment. Subjects were repeatedly roll tilted to angles between 11 and 19 degrees, and then reported their perceived tilt angle using a subjective visual vertical task. They did this while experiencing centripetal acceleration equivalent to Earth gravity (1 Gz), and then hypogravity (0.5 Gz). We hypothesized that, after entering hypogravity, subjects would tend to underestimate their tilt angle. We calculated the percent change in their perception of tilt between 1 Gz and 0.5 Gz.
Time Frame: 1 session
Measure: Mean (Full Range); unit: percentage change
Groups:
- Training, Placebo: placebo
  Hyper gravity training: Subject receives hypergravity training before testing
  Placebo: Placebo
Arm/Group | Training, Placebo
Number analyzed (Participants) | 9
percentage change | 27.0 [7.4 to 57.1]

2. Primary Outcome: Yaw Perceptual Motion Threshold
Description: This is a perceptual self-motion threshold that measures the precision of the vestibular system. It is analogous to an audiogram, but for motion. Subjects sat on a motorized platform which repeatedly provided them with small motions to the left or right. After each motion subjects report whether they perceived a motion to the left or right. Based on subject responses, a psychometric curve fit is performed that determines the threshold (the standard deviation of the underlying cumulative Gaussian). Yaw rotation means rotations about an axis that is perpendicular to gravity.
  This outcome measure applies only to arm 5 subjects.
Time Frame: 2 sessions separated by at least four days; measurements made 2 hrs after ingestion of medication
Measure: Geometric Mean (Standard Deviation); unit: deg per sec
Groups:
- Perceptual Thresholds,Placebo Then Drug: Subjects undergo perceptual motion threshold tests to determine the smallest motion they can reliably sense for yaw rotation, interaural translation and roll tilt. Each subject is tested twice, once with placebo then once with promethazine, separated by >4 days.
Arm/Group | Perceptual Thresholds,Drug Then Placebo | Perceptual Thresholds,Placebo Then Drug
Number analyzed (Participants) | 5 | 5
deg per sec
  Placebo | .83 (.25) | .92 (.29)
  Promethazine | .86 (.19) | 1.06 (.26)

3. Primary Outcome: Roll Perceptual Motion Threshold
Description: This is a perceptual self-motion threshold that measures the precision of the vestibular system. It is analogous to an audiogram, but for motion. Subjects sat on a motorized platform which repeatedly provided them with small motions to the left or right. After each motion subjects report whether they perceived a motion to the left or right. Based on subject responses, a psychometric curve fit is performed that determines the threshold (the standard deviation of the underlying cumulative Gaussian). Roll tilt means rotations about an axis that is Earth-horizontal.
  This outcome measure applies only to arm 5 subjects.
Time Frame: 2 sessions separated by at least four days; measurements made 2 hrs after ingestion of medication
Measure: Geometric Mean (Standard Deviation); unit: deg per sec
Arm/Group | Perceptual Thresholds,Drug Then Placebo | Perceptual Thresholds,Placebo Then Drug
Number analyzed (Participants) | 5 | 5
deg per sec
  Placebo | .27 (.15) | .32 (.12)
  Promethazine | .39 (.20) | .39 (.13)

4. Primary Outcome: Interaural Perceptual Motion Threshold
Description: This is a perceptual self-motion threshold that measures the precision of the vestibular system. It is analogous to an audiogram, but for motion. Subjects sat on a motorized platform which repeatedly provided them with small motions to the left or right. After each motion subjects report whether they perceived a motion to the left or right. Based on subject responses, a psychometric curve fit is performed that determines the threshold (the standard deviation of the underlying cumulative Gaussian). Interaural translation refers to translations in the horizontal plane to the subject's left or right.
  This outcome measure applies only to arm 5 subjects.
Time Frame: 2 sessions separated by at least four days; measurements made 2 hrs after ingestion of medication
Measure: Geometric Mean (Standard Deviation); unit: cm per sec
Arm/Group | Perceptual Thresholds,Drug Then Placebo | Perceptual Thresholds,Placebo Then Drug
Number analyzed (Participants) | 5 | 5
cm per sec
  Placebo | .57 (.17) | .78 (.23)
  Promethazine | .77 (.39) | .80 (.16)

5. Primary Outcome: Percent Change in Manual Control Performance After Exposure to Hypogravity
Description: Note that this applies to arms 6-9 only.
  Subjects sat on a chair on a moving platform on top of a centrifuge that created an artificial gravity environment. Subjects completed a manual control task in which their charge was randomly perturbed in roll tilt, and they used a joystick to attempt to keep themselves aligned with upright, while in the dark. They did this while experiencing centripetal acceleration equivalent to Earth gravity (1 Gz), and then hypogravity (0.5 Gz). We calculated their performance by calculating the standard deviation of chair position across time, with a smaller number indicating better performance. Then we calculated the percent change in their performance between 1 Gz and 0.5 Gz.
Time Frame: 1 session
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Training, Placebo
Number analyzed (Participants) | 10
percentage change | 75.4 (48.8)

ADVERSE EVENTS:
Time Frame: 1 week
Arm/Group | Tilt Perception, Training, Placebo | Tilt Perception, No Training, Placebo | Tilt Perception, Training, Promethazine | Tilt Perception, No Training, Promethazine | Perceptual Threshold Testing: Promethazine | Perceptual Motion Threshold Testing: Placebo | Manual Control, Training, Placebo | Manual Control, No Training, Placebo | Manual Control, Training, Promethazine | Manual Control, No Training, Promethazine
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/0 | 0/0 | 0/0 | 0/10 | 0/10 | 0/10 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/0 | 0/0 | 0/0 | 0/10 | 0/10 | 0/10 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/10 | 0/0 | 0/0 | 0/0 | 0/10 | 0/10 | 0/10 | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No